CLINICAL TRIAL: NCT03580915
Title: Effectiveness of a Functional Literacy Program for Formerly Homeless Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Sharon Gutman, Professor of Rehabilitation and Regenerative Medicine (Occupatio, Rehab & Regenerative Med OT), Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAR8206
Record Dates: First submitted 2018-06-25; First posted 2018-07-10 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Literacy
Keywords: functional literacy; homelessness; daily life activities
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Intervention Model Description: Approximately 10 participants will be randomly assigned to an intervention group; another 10 will be randomly assigned to a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Literacy Intervention (Experimental): The intervention group will receive the functional literacy program in which, in small groups, participants learn literacy skills in the context of daily life activities such as shopping, meal preparation, and transportation use.
  Interventions: Behavioral: Functional Literacy Program; Behavioral: Usual Care Management Services
- Functional Literacy Control (Active Comparator): The control group will not receive intervention but the Usual Care Management Services.
  Interventions: Behavioral: Usual Care Management Services

INTERVENTIONS:
Behavioral: Functional Literacy Program — The intervention will be provided twice weekly in 2-hour sessions, over 8 weeks. The 16 intervention sessions will provide the opportunity for participants to learn functional literacy skills to (1) manage an apartment, (2) access community resources, (3) manage finances, (4) access free recreational activities. All sessions will address literacy skills needed to complete basic daily life activities in the home and community environments. Literacy skills will first be learned and practiced within the supported shelter, and then extended to the community.
  Arms: Functional Literacy Intervention
Behavioral: Usual Care Management Services — The control group will receive the usual housing services without additional intervention.

SUMMARY:
The purpose of this study is to assess a functional literacy program for formerly homeless adults now residing in supported housing who have difficulty performing daily life skills requiring functional literacy (e.g., bill paying, medication management, community transportation) needed to maintain housing placements. The hypothesis is that intervention group participants will improve in functional literacy compared to the control group that does not receive the intervention.

DETAILED DESCRIPTION:
Sixty-five percent of homeless adults are reported to be illiterate or marginally literate. The lack of literacy in a high technological society negatively impacts this population's ability to participate in daily life activities including finding and maintaining employment, renting and maintaining an apartment, seeking health care, using public transportation, and managing finances. Poor literacy marginalizes this population from societal participation and maintains this group in a state of lack and deficiency.

A literacy program will be delivered to participants who are formerly homeless and now residing in supported shelter. Participants will be randomly assigned to an intervention (n=20) or control (n=20) group. The intervention group will receive the functional literacy intervention over 8 weeks, twice weekly. Intervention sessions will allow participants to learn literacy skills within the context of real-life daily activities like grocery shopping, preparing a meal, and purchasing subway cards. Control group participants will not receive intervention.

ELIGIBILITY:
Inclusion Criteria:

* Resident of a supported shelter environment (after homelessness)
* Self-reported difficulty with basic reading skills needed to participate in desired daily life activities
* English-speaking

Exclusion Criteria:

* Severe behavioral management disorder that would make cooperation and direction following problematic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) score | 1-week post-intervention
  The Canadian Occupational Performance Measure (COPM) is a 5-item, 10-point rating scale (1=most important, 10=least important) designed to be completed conjointly by a therapist and participant, and requires approximately 30 minutes to administer. The scale allows participants to identify and prioritize the most important problems impacting daily function and can be used with clients of all ages and diagnoses. Participants are asked to identify the five most critical problems impeding functional performance in the areas of self-care, productivity, and leisure. After the identification of five problems, participants are asked to rate both performance and satisfaction levels of the identified activities on a 10-point scale (1=not satisfied; 10=extremely satisfied). An open-ended narrative section is provided to allow therapists to record participant comments. The COPM is intended to be used pre- and post-intervention.

SECONDARY OUTCOMES:
Inventory of Reading Occupations (IRO) score | 1-week post-intervention
  The IRO-Adult identifies reading materials from a list of 14 categories (e.g., financial records, federal/state aid documents, food and nutrition labels) that participants access as part of daily occupations. Two sections include Reading Categories (having 14 items) and Dimensions of Reading Participation (consisting of 5 dimensions with two open-ended questions and three 5-point Likert scale items; scores of 10+ = higher reading proficiency). For each client-identified reading category, participants are asked a series of questions about the 5 dimensions of reading participation: (1) reading material type; (2) frequency of access; (3) effectiveness, efficiency, and satisfaction; (4) importance of reading material in daily life; and (5) strategies and supports needed to access). The IRO-Adult descriptively assesses participants' relative mastery (effectiveness, efficiency, satisfaction) in functional literacy in relation to occupational participation.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Gutman, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No